CLINICAL TRIAL: NCT02677948
Title: Phase I/II, Open Label, Multicenter Study of Pacritinib Combined With Ibrutinib in Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Brief Title: Multicenter Study of Pacritinib Combined With Ibrutinib in Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: FDA has placed all trials involving Pacritinib on Full Clinical Hold
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2015.131; HUM00105554 (Other: University of Michigan)
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Chronic Lymphocytic Leukemia; Lymphoma, Small Lymphocytic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pacritinib and Ibrutinib (Experimental): Phase I: Patients will receive Pacritinib 100-200 mg twice daily along with Ibrutinib 420mg/day.
  Phase II Lead-In: Pacritinib at MTD daily continuous x 2 months followed by Pacritinib at MTD twice daily along with Ibrutinib 420mg/day.
  Interventions: Drug: Pacritinib; Drug: Ibrutinib

INTERVENTIONS:
Drug: Pacritinib
Drug: Ibrutinib

SUMMARY:
This study combines two drugs in the treatment of relapsed/refractory chronic lymphocytic leukemia (CLL) and small lymphocytic lymphoma (SLL). Investigators are proposing combining ibrutinib, an orally-administered, small molecule inhibitor of Bruton's tyrosine kinase (FDA approved for the treatment of relapsed/refractory CLL), with pacritinib, a novel JAK2-FLT3 inhibitor that has shown activity in relapsed lymphoma, including CLL/SLL. Investigators will first demonstrate the safety and tolerability of Pacritinib when combined with Ibrutinib in a phase I study, which will help establish the MTD (Maximum Tolerated Dose)of Pacritinib when combined with Ibrutinib. Once the optimal dose of Pacritinib is established in the phase I setting, a phase II evaluation will seek to establish the efficacy of the combination of Pacritinib with Ibrutinib. Patients will receive continuous treatment until progressive disease and will be followed while on study treatment for a total of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL/SLL
* Relapsed or refractory CLL or SLL following at least 1 prior line of systemic therapy with active disease meeting criteria for treatment
* Age ≥18 and <80
* ECOG (Eastern Cooperative Oncology Group) ≤2 (This is a performance status that attempts to quantify a patients daily activities where 0 represents normal activity and 5 represents death)
* Adequate organ function defined as AST and ALT ≤ 2 times upper limit of normal (ULN), Total Bilirubin ≤ 1.5 times ULN (exception of Gilbert disease), Renal function: CrCl ≥30 mL/min, Bazett-corrected Q-T interval ≤ 0.45 seconds
* Peripheral blood counts of ANC >500 cells/μL, platelets ≥ 50,000 cells/ μL, Hemoglobin≥ 8 g/dL
* Prior treatment allowed if: at least 30 days have elapsed since last chemotherapy and/or radiation and patient has recovered from all clinically significant treatment-related toxicity, or at least 90 days have passed since date of autologous stem cell transplant and patient has recovered to ≤grade 1 toxicity related to this procedure.
* Ability to provide written informed consent
* Ability to take oral medications.

Exclusion Criteria:

* Pregnant or breast feeding women
* Primary or metastatic CNS (Central Nervous System) disease prior to study enrollment
* Uncontrolled current illness including, but not limited to, ongoing or active infections requiring intravenous antimicrobials, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia and/or psychiatric illness or social situations that would limit compliance with study requirements
* Known HIV infection
* Active infection with Hepatitis B or C virus
* Concomitant therapy in last 30 days of any of the following: cytotoxic chemotherapy, immunosuppressive agents, other investigational therapies or chronic use of systemic corticosteroids
* Prior treatment with ibrutinib
* Uncontrolled autoimmune hemolytic anemia (AIHA) or autoimmune thrombocytopenia (ITP).
* Requires anticoagulation with warfarin or equivalent Vit K antagonist
* Allergy to either ibrutinib or pacritinib or components within medication
* Treatment with strong CYP3A4 inducer or inhibitor, for which no alternative is available.
* Unwilling or unable to use a medically acceptable form of contraception.
* Any gastrointestinal or metabolic condition that could interfere with the absorption of oral medication.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Then maximum tolerated dose (MTD) of Pacritinib when given in combination with Ibrutinib | 28 Days
  DLTs (Dose Limiting Toxicities) occurring during the 1st cycle (first 28 days) of treatment with the combination of pacritinib and ibrutinib will be used for dose-escalation decisions. MTD is defined as the largest dose at which no more than 25% of patients experience a DLT.
The number of patients with a Complete Response (CR) | 2 Years Post Treatment
  Patients will be followed for response from the date of initial treatment until 2 years post treatment. CR is defined as:
  Lymphadenopathy - None ˃1.5 cm Hepatomegaly - None Splenomegaly - None Blood Lymphocytes - ˂ 4000/μL Bone Marrow - Normocellular, 30% lymphocytes, no B-lymphoid nodules. Platelet Count - ˃ 100,000/μL Hemoglobin - ˃ 11.0 g/dL Neutrophils - ˃ 1,500/μL

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Wilcox, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota